CLINICAL TRIAL: NCT04363944
Title: A Functional Upper Limb Training and Assessment Tool to Enhance Efficacy and Scalability of Rehabilitation in Ecological Environments
Brief Title: Smartphone and 3D Printing Based Home Rehabilitation System for Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeanne Langan, Principal Investigator, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 78849; 1R21HD092243 (NIH)
Record Dates: First submitted 2020-04-16; First posted 2020-04-27 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: home programs; assistive technology; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The purpose of the intervention was to provide proof of concept that it is feasible for individuals with stroke to use mRehab in a home program and to examine if changes in motor function were enhanced following the home program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mRehab (Experimental): Use of mRehab in a home program completing unilateral and bilateral activities. Participants are able to complete unilateral activities with their paretic arm/hand
  Interventions: Device: mRehab
- mRehab completing all activities bilaterally (Experimental): Use of mRehab in a home program completing unilateral and bilateral activities. Participantsare can only complete intended unilateral activities using both hands
  Interventions: Device: mRehab

INTERVENTIONS:
Device: mRehab — mRehab (mobile Rehab) was created to better support in-home upper limb rehabilitation programs. It incorporates a task-oriented approach and immediate performance-based feedback. mRehab consists of 3D-printed household items (a mug, bowl, key, and doorknob) integrated with a smartphone and an app. The app guides participants through practice of activities of daily living (ADL), for example, sipping from a mug. It can also consistently measure time to complete an activity and quality of movement (smoothness/accuracy) during the performance of ADLs. In each session of exercise participants receive feedback on the number of repetitions they complete for each activity, the average time to complete the activity and the average smoothness to perform the activity. Participants were trained in use of mRehab in lab visits and then took mRehab home to use the system. mRehab recorded longitudinal data.

SUMMARY:
Interventions promoting optimum motor performance across the lifespan are a priority after a neurological insult such as stroke. The proposed research incorporates smart devices and 3D printing to create a patient-centered rehabilitation device, mRehab. This innovative blend of technology and principles of neuroplasticity can advance standards of practice in healthcare. In this feasibility study, it is hypothesized that individuals with chronic stroke can successfully use the portable rehabilitation unit, mRehab, at home with minimal oversight from the research team. Use of mRehab in a home based setting and functional changes in upper limb movement will be assessed.

DETAILED DESCRIPTION:
Impairments following stroke make it one of the leading causes of disability. Many individuals with stroke do not recover complete function of the upper limb at time of discharge from clinical services. Moreover, early stage improvements may wane following the cessation of formal therapies. Regaining as much upper limb function as possible is important, as even mild impairments are associated with limitations in daily function and lower health-related quality of life. The overarching purpose of this project is to use portable technology, affordable for home use, to provide objective feedback on performance of upper limb motor tasks to individuals with residual deficits following chronic conditions such as stroke. Objective feedback serves to better inform the participant of their progress and actively engage them in their rehabilitation, thus encouraging self-management of rehabilitation. Results from a recent survey shows therapists predominantly provide patients with stroke written home exercise programs at time of discharge from therapies. With this static approach, patients have a limited capacity to evaluate their motor performance and no encouragement to refine their movement. Smartphones were coupled with three-dimensional (3D) printed objects to create a home rehabilitation system, mRehab. The built-in sensors in smartphones and a custom app can quantify characteristics of movement and provide actionable feedback to users during in-home rehabilitation. It was hypothesized that 1) participants with stroke could use mRehab in a home program with minimal oversight and 2) use of mRehab would result in changes in functional movement.

Methodology: A single-subject experimental design with multiple baselines was used. A strength of the single-subject study design is that participants serve as their own control. Each participant had a varying length of the baseline and follow-up periods to establish that the intervention, rather than time, was the primary reason for any observed change in performance. Participants completed baseline measurements, a six-week mRehab home program, and follow-up measurements. Baseline measurements consisted of both in-lab and in-home measurements. Participants attended two lab visits prior to starting the home program to establish baselines on clinical assessments and to learn how to use mRehab. MRehab collected limited preliminary performance data without providing feedback during baseline. Participants then used mRehab in a six week home program receiving feedback on their performance each time they completed practice of an activity. At the completion of the home program participants completed follow up assessments that were similar to the baseline measurements. In addition, usability of mRehab was assessed.

ELIGIBILITY:
Individuals in the intervention all had a history of stroke.

Inclusion Criteria for feasibility study:

1. at least 18 years of age and living in the community
2. had a history of one stroke six or more months previous
3. had a minimum score of 124 on the Mattis Dementia Rating Scale (MDRS).

Exclusion Criteria for feasibility study:

1. acute or chronic pain that would interfere with participation
2. severely limited range of motion or contractures of shoulder, elbow, wrist or hand,
3. absent or severely impaired proprioception of the upper limb
4. musculoskeletal or circulatory conditions affecting the upper limb such as vascular disease, tendonitis, cellulitis, Raynaud's syndrome, or severe osteoarthritis or rheumatoid arthritis
5. spasticity graded as 3 or greater for upper extremity movement on the Modified Ashworth Scale (MAS)
6. botulinum toxin injections for spasticity management within three months of starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Langan, PT, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic information (such as age and gender) cognitive assessments, motor performance on clinical assessments and data collected during rehabilitation from mRehab.
Time Frame: The IPD will be provided following acceptance of manuscripts.
Access Criteria: Individual participant data (IPD) will be provided for the primary and secondary outcomes of the study. Data will be available in June 2022 and will continue to be available for 2 years, June 2024. The IPD may be accessed by the URL: https://cse.buffalo.edu/~wenyaoxu/project/mRehab_Data.xlsx
URL: https://cse.buffalo.edu/~wenyaoxu/project/mRehab_Data.xlsx

REFERENCES:
- [Derived] Bhattacharjya S, Cavuoto LA, Reilly B, Xu W, Subryan H, Langan J. Usability, Usefulness, and Acceptance of a Novel, Portable Rehabilitation System (mRehab) Using Smartphone and 3D Printing Technology: Mixed Methods Study. JMIR Hum Factors. 2021 Mar 22;8(1):e21312. doi: 10.2196/21312. PMID 33749608
- [Derived] Langan J, Bhattacharjya S, Subryan H, Xu W, Chen B, Li Z, Cavuoto L. In-Home Rehabilitation Using a Smartphone App Coupled With 3D Printed Functional Objects: Single-Subject Design Study. JMIR Mhealth Uhealth. 2020 Jul 22;8(7):e19582. doi: 10.2196/19582. PMID 32706702

RESULTS

PARTICIPANT FLOW:
Groups:
- Use of mRehab in a Home Program: mRehab incorporates a task-oriented approach and immediate performance-based feedback and longitudinal data. mRehab consists of 3D-printed household items integrated with a smartphone and an app that guides participants through practice of ADLs.
  Single subject design with varying lengths of baseline data acquisition and follow-up data acquisition 2 visits to establish baseline Intervention: 6-week in home training program using mRehab 2 visits to establish performance immediately following intervention and 1-3 weeks post. Participants that completed baseline data acquisition, training and follow up were included in the final analyses. If a participant used hand over hand to complete all mrehab activities. Their data was not included in the analyses.
- Use of mRehab in Home Completing All Activities Bilaterally: Participant completed all activities in the six week in home mRehab program bilaterally.
Period: Overall Study
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in Home Completing All Activities Bilaterally
Started | 18 | 1
Completed | 16 | 1
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Individuals with stroke that completed baseline analyses and completed all assessments and training unilaterally with their paretic hand/arm.
Groups:
- Use of mRehab in a Home Program: mRehab incorporates a task-oriented approach and immediate performance-based feedback. mRehab consists of 3D-printed household items integrated with a smartphone and an app. The app guides participants through practice of activities of daily living. In each session of exercise participants receive feedback on the number of repetitions they complete for each activity, the average time to complete the activity and the average smoothness to perform the activity. Participants were trained in use of mRehab in lab visits and then took mRehab home to use the system. mRehab recorded longitudinal data. Participants included in this group demonstrate the ability to complete mRehab tasks unilaterally.
- Use of mRehab in a Home Program Completing All Activities Bilaterally: Participant completed all activities in data collection and in the six week in home mRehab program bilaterally.
- Total: Total of all reporting groups
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in a Home Program Completing All Activities Bilaterally | Total
Number analyzed (Participants) | 16 | 1 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.82 (13.22) | 22 | 60.32 (15.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 10 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 1 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 1 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 1 | 17
Time to complete activity in the mRehab home program [Mean (Standard Deviation); unit: seconds] — The average time to complete an activity in mRehab on day 1 of the 6 week home program.
  seconds
    Vertical bowl transfer | 5.04 (.91) | 6.63 | 5.13 (.97)
    Horizontal bowl transfer | 5.03 (1.32) | 4.87 | 5.02 (1.28)
    Vertical mug transfer | 5.22 (1.22) | 5.39 | 5.23 (1.09)
    Horizontal mug transfer | 4.96 (1.22) | 5.19 | 4.97 (1.18)
    Simulate sip from mug | 9.51 (4.71) | 9.38 | 9.50 (4.64)
    Enter phone number | 30.86 (26.28) | 38.22 | 31.29 (25.50)
    quick tap | 17.05 (9.42) | 8.78 | 16.56 (9.34)
Average smoothness per activity in the mRehab home program [Mean (Standard Deviation); unit: jerk score] — The average smoothness per activity in mRehab on the first day of the 6 week home program.
  Using the acceleration readings from the inertial measurement unit in the smartphone, a normalized jerk score which is dimensionless, allowing comparisons of movements that vary in duration and/or amplitude, can be computed. There are no set upper bounds, as the score is dependent on the smoothness. The minimum score is 0, which would indicate no jerk, or perfectly smooth movement. The score provides relative information for each movement, a normal range has not been established for each movement.
  jerk score
    Vertical bowl transfer | 511.99 (297.33) | 1727.74 | 583.51 (412.10)
    Horizontal bowl transfer | 478.53 (315.49) | 1015.74 | 510.13 (332.1)
    Vertical mug transfer | 699.24 (321.74) | 1254.94 | 731.93 (339.46)
    Horizontal mug transfer | 585.83 (233.81) | 485.56 | 579.93 (227.69)
    Simulate sip from mug | 394.17 (239.46) | 385 | 393.63 (231.86)
Wolf Motor Function Test- Ave time to complete a task over 2 testing sessions using the WMFM [Mean (Standard Deviation); unit: seconds] — The Wolf Motor Function Test (WMFT) is used to assess function of the upper extremity. The 17 item version of the WMFT was used. Tasks in the WMFT include tasks that assess gross motor activity (such as lifting hand/arm and placing it on a box), fine motor activity (such as picking up a paper clip) and strength. One timed task is a bilateral task (folding a towel). For timed tasks, participants are given up to 120 seconds to complete the task. If they cannot successfully complete it in that time they are given the max score of 120 seconds. We report the average time to complete an activity.
  seconds | 17.62 (22.16) | 96.28 (0) | 19.90 (27.96)
Nine hole peg test average time to complete over 2 testing sessions [Mean (Standard Deviation); unit: seconds] — The participant places 9 pegs into 9 holes and then removes the pegs. The stop watch is started when the patient touches the first peg and stopped when the patient takes out the last peg from the peg hole and places the it in the container. If participants were unable to complete the task of placing all 9 pegs in a hole, they were given a score of 300 seconds.
  seconds | 135.52 (115.91) | 300 (0) | 144.18 (118.79)

OUTCOME MEASURES:

1. Primary Outcome: Repetitions Completed for Each Activity in the mRehab Home Program
Description: The total number of repetitions each participant completed for each activity in mRehab during the 6 week home program was recorded. The average total number of repetitions completed for each activity is reported.
Time Frame: 6 week in-home program
Population: 16 participants with chronic stroke that completed mRehab in-home training with their paretic hand.
Measure: Mean (Standard Deviation); unit: repetitions
Groups:
- Use of mRehab in a Home Program: mRehab incorporates a task-oriented approach and immediate performance-based feedback. mRehab consists of 3D-printed household items integrated with a smartphone and an app. The app guides participants through practice of activities of daily living. In each session of exercise participants receive feedback on the number of repetitions they complete for each activity, the average time to complete the activity and the average smoothness to perform the activity. Participants were trained in use of mRehab in lab visits and then took mRehab home to use the system. mRehab recorded longitudinal data.
  * Participants that met inclusion/exclusion criteria n=19
  * Participants that completed baseline data acquisition, training and follow up n=17
    * 1 participant withdrew from study prior to home training citing they did not have sufficient time in their schedule to participate.
    * 1 participant withdrew during the intervention. Participant felt that their caregiver needed to help with the home program and their schedules did not align well to complete the home program
  * Participants included in the analyses n=16
    * 1 participant performed mRehab activities hand over hand using assisting the paretic hand. This participant was not considered part of the group that performed all training unilaterally. Their data is not reported.
- Use of mRehab in a Home Program Completing All Activities Bilaterally: Participant completed all activities in data collection and in the six week in-home mRehab program bilaterally.
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in a Home Program Completing All Activities Bilaterally
Number analyzed (Participants) | 16 | 1
repetitions
  Vertical bowl transfer | 282.06 (210.00) | NA — Home program data was not obtained from smartphone.
  Horizontal bowl transfer | 289.44 (223.34) | NA — Home program data was not obtained from smartphone.
  Vertical mug transfer | 283.69 (227.94) | NA — Home program data was not obtained from smartphone.
  Horizontal mug transfer | 292.31 (224.02) | NA — Home program data was not obtained from smartphone.
  Simulate sip from mug | 202.19 (151.48) | NA — Home program data was not obtained from smartphone.
  Enter phone number | 153.13 (131.05) | NA — Home program data was not obtained from smartphone.
  Quick tap | 177.20 (141.26) | NA — Home program data was not obtained from smartphone.

2. Primary Outcome: Time to Complete Activity in the mRehab Home Program
Description: average time to complete an activity in the mRehab home program
Time Frame: last day of the 6 week in home program
Population: Participants with chronic stroke that completed the mRehab training using their paretic hand.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in a Home Program Completing All Activities Bilaterally
Number analyzed (Participants) | 16 | 1
seconds
  Vertical bowl transfer | 4.03 (.46) | 4.17
  Horizontal bowl transfer | 4.01 (.60) | 4.71
  Vertical mug transfer | 5.22 (1.22) | 9.28
  Horizontal mug transfer | 4.00 (.58) | 4.69
  Simulate sip from mug | 9.62 (1.39) | 9.33
  Enter phone number | 22.35 (14.05) | 25.53
  Quick tap | 14.75 (7.54) | 8.76
Statistical Analysis 1: Comparison: Use of mRehab in a Home Program; mRehab task vertical bowl transfer- moving the bowl vertically up and down; Test type: Equivalence — A paired-t test comparing performance of vertical bowl transfer at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p < 0.001, t-test, 2 sided — Comparing the change in performing a vertical bowl transfer, the calculated p-value for this activity was <.001
Statistical Analysis 2: Comparison: Use of mRehab in a Home Program; mRehab task horizontal bowl transfer- moving the bowl horizontally; Test type: Equivalence — A paired-t test comparing performance of moving the bowl horizontally at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .001, t-test, 2 sided — Comparing the change in performing a horizontal bowl transfer, the calculated p-value for this activity was .001
Statistical Analysis 3: Comparison: Use of mRehab in a Home Program; mRehab task vertical mug transfer- moving the mug vertically up and down; Test type: Equivalence — A paired-t test comparing performance of the vertical mug transfer at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .003, t-test, 2 sided — Comparing the change in performing a vertical mug transfer, the calculated p-value for this activity was .003
Statistical Analysis 4: Comparison: Use of mRehab in a Home Program; mRehab task horizontal mug transfer- moving the mug horizontally; Test type: Equivalence — A paired-t test comparing performance of the horizontal mug transfer at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .009, t-test, 2 sided — Comparing the change in performing a horizontal mug transfer, the calculated p-value for this activity was .009
Statistical Analysis 5: Comparison: Use of mRehab in a Home Program; mRehab task simulate sip- bring mug within one inch of mouth as if taking a drink; Test type: Equivalence — A paired-t test comparing performance of the simulated sip at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .933, t-test, 2 sided; A paired-t test comparing performance at the beginning of the 6 week in-home program to the end of the 6 week in-home program
Statistical Analysis 6: Comparison: Use of mRehab in a Home Program; mRehab task enter phone number; Test type: Equivalence — A paired-t test comparing performance of entering a phone number at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .136, t-test, 2 sided
Statistical Analysis 7: Comparison: Use of mRehab in a Home Program; mRehab task quick tap- tapping a moving object on the phone screen; Test type: Equivalence — A paired-t test comparing performance of the quick tap at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .005, t-test, 2 sided

3. Primary Outcome: Average Smoothness Per Activity in the mRehab Home Program
Description: The average smoothness per activity in mRehab on the first day of the 6 week home program. Using the acceleration readings from the inertial measurement unit embedded in the smartphone, a normalized jerk score which is dimensionless, allowing comparisons of movements that vary in duration and/or amplitude, can be computed. There are no set upper bounds for the score, as it is dependent on the smoothness. The minimum score is 0, which would indicate no jerk, or perfectly smooth movement. This measurement provides relative information for each movement as a normal range has not been established for each of the movements in this study. Overall, a lower score indicates smoother movement.
Time Frame: last day of the 6 week in-home program
Population: 16 participants with chronic stroke performing the in-home rehabilitation unilaterally
Measure: Mean (Standard Deviation); unit: jerk score
Groups:
- Use of mRehab in a Home Program: mRehab incorporates a task-oriented approach and immediate performance-based feedback. mRehab consists of 3D-printed household items integrated with a smartphone and an app. The app guides participants through practice of activities of daily living. In each session of exercise participants receive feedback on the number of repetitions they complete for each activity, the average time to complete the activity and the average smoothness to perform the activity. Participants were trained in use of mRehab in lab visits and then took mRehab home to use the system. mRehab recorded longitudinal data.
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in a Home Program Completing All Activities Bilaterally
Number analyzed (Participants) | 16 | 1
jerk score
  Vertical bowl transfer | 410.66 (128.81) | 768.17
  Horizontal bowl transfer | 375.39 (137.23) | 732.16
  Vertical mug transfer | 492.70 (226.60) | 1869.6
  Horizontal mug transfer | 431.23 (159.97) | 531.8
  simulating sipping from mug | 331.11 (61.77) | 347.17
Statistical Analysis 1: Comparison: Use of mRehab in a Home Program; mRehab task vertical bowl transfer- moving bowl vertically up and down; Test type: Equivalence — Paired t-tests comparing performance at the first session of in-home training to the last session of in-home training were conducted; p = .228, t-test, 2 sided
Statistical Analysis 2: Comparison: Use of mRehab in a Home Program; mRehab task horizontal bowl- bowl moved horizontally; Test type: Equivalence — A paired-t test comparing performance at the beginning of the 6 week in-home program to the end of the 6 week in-home program; p = .196, t-test, 2 sided
Statistical Analysis 3: Comparison: Use of mRehab in a Home Program; mRehab task Vertical Mug- Mug moved vertically and then placed on counter; Test type: Equivalence — [test comment as in outcome 3, analysis 2]; p = .024, t-test, 2 sided
Statistical Analysis 4: Comparison: Use of mRehab in a Home Program; mRehab task horizontal mug transfer- moving the mug horizontally; Test type: Equivalence — [test comment as in outcome 3, analysis 2]; p = .038, t-test, 2 sided
Statistical Analysis 5: Comparison: Use of mRehab in a Home Program; mRehab task simulate sip; Test type: Equivalence — [test comment as in outcome 3, analysis 2]; p = .306, t-test, 2 sided — calculated p-value greater than .05

4. Secondary Outcome: Wolf Motor Function Test
Description: The Wolf Motor Function Test (WMFT) is used to assess function of the upper extremity. The 17 item version of the WMFT was used. Tasks in the WMFT include tasks that assess gross motor activity (such as lifting hand/arm and placing it on a box), fine motor activity (such as picking up a paper clip) and strength. One timed task is a bilateral task (folding a towel). For timed tasks, participants are given up to 120 seconds to complete the task. If they cannot successfully complete it in that time they are given the max score of 120 seconds. In our papers we only use the timed tasks in the WMFT in our analyses. We report the average time to complete a task in the WMFT. A lower score indicates less time is required to complete the task.
Time Frame: within 1 week of the completion of the in-home program
Population: Participants with chronic stroke that performed mRehab activities unilaterally.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in a Home Program Completing All Activities Bilaterally
Number analyzed (Participants) | 16 | 1
seconds | 15.25 (21.31) | 96.27
Statistical Analysis 1: Comparison: Use of mRehab in a Home Program; Test type: Equivalence — The average of the WMFT from testing sessions pre intervention (week 1 and approximately week 2) was compared to the WMFT immediately following mRehab home intervention (week 8) using a two tailed paired t-test; p = .017, t-test, 2 sided — calculated p-value .017

5. Secondary Outcome: Nine Hole Peg Test
Description: A timed clinical assessment used to measure finger dexterity. Lower times represent better performance. Participants place 9 pegs in 9 holes and then remove the pegs and place them in a container. The stop watch starts when the participant touches the first peg and stops when they place the last peg in the container. If participants could not complete placing the pegs in the holes they were given a score of 300 seconds.
Time Frame: within 1 week of the end of the in-home program
Population: Participants with stroke that participated in a home rehabilitation program using mRehab.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- mRehab: Use of mRehab in a home program
  mRehab: mRehab (mobile Rehab) was created to better support in-home upper limb rehabilitation programs. It incorporates a task-oriented approach and immediate performance-based feedback. mRehab consists of 3D-printed household items (a mug, bowl, key, and doorknob) integrated with a smartphone and an app. The app guides participants through practice of activities of daily living (ADL), for example, sipping from a mug. It can also consistently measure time to complete an activity and quality of movement (smoothness/accuracy) during the performance of ADLs. In each session of exercise participants receive feedback on the number of repetitions they complete for each activity, the average time to complete the activity and the average smoothness to perform the activity. Participants were trained in use of mRehab in lab visits and then took mRehab home to use the system. mRehab recorded longitudinal data.
- Use of mRehab at Home Completing Activities Bilaterally: Participant completed all activities in data collection and in the six week in home mRehab program bilaterally.
Arm/Group | mRehab | Use of mRehab at Home Completing Activities Bilaterally
Number analyzed (Participants) | 16 | 1
seconds | 136.36 (108.96) | 300
Statistical Analysis 1: Comparison: mRehab; Compared pre and post intervention data for participants using mRehab for a 6 week home program; Test type: Equivalence — Test, the scores from the first and second in-laboratory visits were averaged to account for variability in the performance of individuals with stroke. This averaged preintervention score was compared with the third in-laboratory visit to assess the immediate change in performance following use of mRehab; p = .019, t-test, 2 sided

6. Secondary Outcome: Difficulty Rating Scale
Description: A scale used to elicit user opinions on ease of use of the 3D printed objects (mug, bowl, key, and doorknob). It was a 7 point likert scale ranging from Very Difficult to Very Easy. The range was -3 to 3. A score of -3 represented the three-dimensional printed object was very difficult to use and a score of 3 representing the object was easy to use. The scores for the mug, bowl, key and door knob are included in the mean score given below.
Time Frame: within 1 - 3 weeks of the end of the program
Population: Participants with stroke that participated in a 6 week home program using mRehab.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Use of mRehab in a Home Program: mRehab incorporates a task-oriented approach and immediate performance-based feedback and longitudinal data. mRehab consists of 3D-printed household items integrated with a smartphone and an app that guides participants through practice of ADLs.
  Single subject design with varying lengths of baseline data acquisition and follow-up data acquisition 2 visits to establish baseline Intervention: 6-week in home training program using mRehab 2 visits to establish performance immediately following intervention and 1-3 weeks post.
Arm/Group | Use of mRehab in a Home Program
Number analyzed (Participants) | 12
units on a scale | 1.07 (1.07)

7. Secondary Outcome: Systems Usability Scale (SUS)
Description: A reliable tool for measuring usability. The Systems Usability Scale (SUS) consists of 10 questions, each rated on a 5-point Likert scale ranging from Strongly agree to Strongly disagree. The SUS was used to assess the participant's satisfaction with the mRehab system. A higher score represents a more positive perception of the device. A score of 50 would represent the strongest agreement that mRehab is a usable system. A score of 10 would represent the strongest disagreement that mRehab is a usable system.
Time Frame: within 1-3 weeks of completion of home program
Population: Participants with stroke that completed a 6 week home program using mRehab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Use of mRehab in a Home Program
Number analyzed (Participants) | 16
units on a scale | 31.25 (3.80)

8. Secondary Outcome: mRehab Acceptance Questionnaire
Description: The mRehab (mobile Rehab) acceptance questionnaire was designed to assess the participants perception of the mRehab system we designed for this study. The questionnaire is based upon the Technology Acceptance model using a seven-point Likert scale - highly disagree (1) to highly agree (7)- for each question. Participants responded to 16 questions that probed the user's perceception of how they interacted with technology (3 questions) and their perceived usefulness, perceived ease of use, and behavioral intention to use the mRehab system in the future (13 questions). The total score is calculated as the sum of the response to each question. A score demonstrating the participant highly agreed that they would interact with technology and that they found mRehab useful, easy to use and that they would use in in the future would be 112. The minimum total score would be 16 (with a rating of highly disagree for each question). Higher scores would indicate better acceptance/interaction.
Time Frame: within 1-3 weeks of completion of the 6 week in-home program
Population: Participants with stroke that used mRehab in a 6 week home program.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Use of mRehab in Home Completing Activities Bilaterally: Participant completed all activities in data collection and in the six week in home mRehab program bilaterally.
Arm/Group | Use of mRehab in a Home Program | Use of mRehab in Home Completing Activities Bilaterally
Number analyzed (Participants) | 16 | 1
units on a scale | 91.56 (11.79) | 106

ADVERSE EVENTS:
Time Frame: 10 weeks including in-lab pre-test, 6 week in-home program, and in-lab post-test
Description: Adverse events were monitored, but none were reported/ observed.
Groups:
- Use of mRehab in a Home Program: mRehab incorporates a task-oriented approach and immediate performance-based feedback and longitudinal data. mRehab consists of 3D-printed household items integrated with a smartphone and an app that guides participants through practice of ADLs. Individuals that completed all outcome measures unilaterally with their paretic arm/hand were included in this group.
  Single subject design with varying lengths of baseline data acquisition and follow-up data acquisition 2 visits to establish baseline Intervention: 6-week in home training program using mRehab 2 visits to establish performance immediately following intervention and 1-3 weeks post.
  In total, it took 10 weeks for participants to complete the study.
Arm/Group | Use of mRehab in a Home Program
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04363944/Prot_SAP_000.pdf